CLINICAL TRIAL: NCT01907412
Title: Trial of Transition to Parenthood Program for Couples
Acronym: FF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Mark Feinberg, Research professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD058529-02 (NIH)
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Parent-Child Relations
Keywords: First time parents; Coparenting; Family Foundations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Couples in the Control group did not receive the Family Foundations Coparenting Program.
- Intervention Group (Experimental): Couples randomly assigned to the Intervention Group received the Family Foundations Coparenting Program.
  Interventions: Behavioral: Family Foundations Coparenting Program

INTERVENTIONS:
Behavioral: Family Foundations Coparenting Program — Family Foundations, a program for adult couples expecting their first child, is designed to help them establish positive parenting skills and adjust to the physical, social, and emotional challenges of parenthood. Program topics include coping with postpartum depression and stress, creating a caring environment, and developing the child's social and emotional competence.
  Family Foundations is delivered to groups of couples through four prenatal and four postnatal classes of 2 hours each. Prenatal classes are started during the fifth or sixth month of pregnancy, and the postnatal classes end when the children are 6 months old.
  Family Foundations is delivered in a community setting by childbirth educators who have received 3 days of training from Family Foundations staff.
  Arms: Intervention Group

SUMMARY:
This is a research study to evaluate the effectiveness of the Family Foundations program and to better understand how families cope with having a new baby. The research questions include: What is the effectiveness of the Family Foundations program? How do families cope with having a new baby?

ELIGIBILITY:
Inclusion Criteria:

* Expecting first child
* Couple living together and planning to raise child together
* 18 years or older

Exclusion Criteria:

* not first child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2008-06; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Coparenting Quality | Up to 2.5 years from baseline
  We assessed coparenting relationship quality with the 31-item Coparenting Scale, which was created based on prior work (e.g., Abidin & Brunner, 1995; Cordova, 2001; Frank, Olmstead, Wagner,& Laub, 1991; Margolin et al., 2001; McHale, 1997). The overall score represents an average of items covering theoretically important domains: coparental agreement, support,undermining, and exposure of the child to conflict.

SECONDARY OUTCOMES:
Aggressive Parenting | Up to 2.5 years after baseline
  Aggressive parenting was measured using Parent-Child Conflict Tactics Scales (Straus et al., 1998).

OTHER OUTCOMES:
Cardiovascular disease risk | 8 years from baseline
  We assessed parent and child cardiovascular disease risk via inflammatory (C-reactive protein, Interleukin-6) and metabolic (total cholesterol, glycated hemoglobin, body mass index, blood pressure) outcomes previously linked to cardiovascular disease risk (e.g., Danesh et al., 2004; Goran et al., 2003; Ortega et al., 2016; Fuchs et al., 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, Prevention Research Center, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Aytuglu A, Graham-Engeland JE, Feinberg ME, Murray-Perdue SA, Conway CA, Schreier HMC. Longitudinal associations between father- and mother-child interactions, coparenting, and child cardiometabolic health. Health Psychol. 2025 Dec 1:10.1037/hea0001567. doi: 10.1037/hea0001567. Online ahead of print. PMID 41325157
- [Derived] Aytuglu A, Graham-Engeland JE, Feinberg ME, Jones DE, Schreier HMC. Child sleep problems mediate prospective associations between fathers' parenting stress and child blood glucose levels. J Fam Psychol. 2025 Mar;39(2):277-283. doi: 10.1037/fam0001306. Epub 2025 Jan 16. PMID 39818869
- [Derived] Schreier HMC, Feinberg ME, Jones DE, Ganguli A, Givens C, Graham-Engeland J. Children's empathy moderates the association between perceived interparental conflict and child health. Brain Behav Immun. 2024 May;118:128-135. doi: 10.1016/j.bbi.2024.02.022. Epub 2024 Feb 24. PMID 38408496
- [Derived] Jones EJ, Feinberg ME, Graham-Engeland JE, Jones DE, Schreier HMC. A perinatal coparenting intervention: Effects of a randomized trial on parent cardiometabolic risk and self-reported health. Biol Psychol. 2023 Oct;183:108664. doi: 10.1016/j.biopsycho.2023.108664. Epub 2023 Aug 23. PMID 37625684
- [Derived] Feinberg ME, Jones DE, Roettger ME, Hostetler ML, Sakuma KL, Paul IM, Ehrenthal DB. Preventive Effects on Birth Outcomes: Buffering Impact of Maternal Stress, Depression, and Anxiety. Matern Child Health J. 2016 Jan;20(1):56-65. doi: 10.1007/s10995-015-1801-3. PMID 26194453